CLINICAL TRIAL: NCT00053573
Title: An Open-Label, Multicenter, Multinational, Study of the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of rhGAA Treatment in Patients Greater Than 6 Months and Less Than or Equal to 36 Months Old With Infantile-Onset GSD-II
Brief Title: rhGAA in Patients With Infantile-onset Glycogen Storage Disease-II (Pompe Disease)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU01702
Record Dates: First submitted 2003-01-31; First posted 2003-02-03 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Glycogen Storage Disease Type II; Pompe Disease; Acid Maltase Deficiency Disease; Glycogenosis 2
Keywords: Glycogen Storage Disease Type II; GSD-II; Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Myozyme

INTERVENTIONS:
Biological: Myozyme — 20 mg/kg to 40 mg/kg qow
  Other Names: Alglucosidase alfa

SUMMARY:
Glycogen Storage Disease Type II ("GSD-II"; also known as Pompe disease) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with GSD-II, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. This study is being conducted to evaluate the safety and effectiveness of recombinant human acid alpha-glucosidase (rhGAA) as a potential enzyme replacement therapy for GSD-II. Patients diagnosed with infantile-onset GSD-II who are greater than 6 months old, but less than or equal to 36 months old will be studied.

ELIGIBILITY:
Inclusion Criteria:

* The patient or the patient's legal guardian(s) must provide written informed consent prior to any study-related procedures being performed
* The patient must have a clinical diagnosis of infantile GSD-II as defined by: (a) the patient has/had documented (in a medical record) onset of symptoms compatible with GSD-II by 12 months of age; (b) the patient has documented GAA deficiency as illustrated by an endogenous GAA activity less than or equal to 2% of the mean of the normal range as assessed in cultured skin fibroblasts; AND (c) the patient has a Left Ventricular Mass Index greater than 2 standard deviations above the mean for age
* The patient is greater than 6 months old and less than or equal to 36 months old at the time of the first dose of rhGAA
* The patient and his/her legal guardian(s) must have the ability to comply with the clinical protocol

Exclusion Criteria:

* Signs and symptoms of cardiac failure and an ejection fraction less than 40%
* Major congenital abnormality
* Clinically significant organic disease (with the exception of symptoms relating to GSD-II), including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial or potentially decrease survival
* Use of any investigational product within 30 days prior to study enrollment
* Received enzyme replacement therapy with GAA from any source

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2003-02; Primary Completion 2006-07 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of Myozyme | 52 weeks
Determine proportion of patients alive over the course of treatment | 52 weeks
PK profile of MZ | 52 weeks
PD profile of MZ | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- United States (3):
  - University of Florida College of Medicine, Gainesville, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
- Pediatrique Hopital de Brousse, Lyon, France
- Rambam Medical Center, Haifa, Israel
- Royal Manchester Children's Hospital, Manchester, United Kingdom

REFERENCES:
- [Derived] Kishnani PS, Goldenberg PC, DeArmey SL, Heller J, Benjamin D, Young S, Bali D, Smith SA, Li JS, Mandel H, Koeberl D, Rosenberg A, Chen YT. Cross-reactive immunologic material status affects treatment outcomes in Pompe disease infants. Mol Genet Metab. 2010 Jan;99(1):26-33. doi: 10.1016/j.ymgme.2009.08.003. PMID 19775921